CLINICAL TRIAL: NCT01755390
Title: A Phase I Dose Finding Study of XRP6258 Administered as a Weekly 1-hour Intravenous Infusion to Patients With Advanced Solid Tumors
Brief Title: A Dose Finding Study of XRP6258 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED6189
Record Dates: First submitted 2012-12-17; First posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): IV escalation part:
  XRP6258 administered as a 1-hour IV infusion on Days 1, 8, 15 and 22 of each 5-week cycle until evidence of disease progression, unacceptable toxicity or patient's withdrawal.
  Oral bioavailability part:
  XRP6258 administered at the dose of 8.4 mg/m² as an oral administration on Day 1 Cycle 1 and as a weekly 1-hour i.v. infusion at the subsequent weeks of treatment. Patients receiving oral administration at Day 1, Cycle 1 are to fast for 12 hours before and 4 hours after administration.
  Interventions: Drug: Cabazitaxel (XRP6258)

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form: infusion solution Route of administration: Intravenous
  Other Names: Jevtana

SUMMARY:
Primary Objective:

- To determine the maximum tolerated dose (MTD) and the dose-limiting toxicity (DLT) of XRP6258 when given as a weekly 1-hour intravenous (i.v.) infusion for the first 4 consecutive weeks of each 5-week treatment cycle (Day 1, Day 8, Day 15, Day 22 of each 5-week treatment cycle).

Secondary Objectives :

* To define the safety profile of the drug
* To establish the recommended dose and time interval for future Phase II trials
* To determine the pharmacokinetic (PK) profile of XRP6258 in man
* To assess the absolute oral bioavailability of XRP6258 at the i.v. recommended dose (following Protocol Amendment No. 2)
* To look for evidence of antitumor activity

DETAILED DESCRIPTION:
The duration of the study will include the following periods:

* Pretreatment: 28 to 7 days before first infusion
* Treatment: Weekly for the first four consecutive weeks during 5-week treatment cycle
* Post-treatment: 3 - 4 weeks after last infusion.

Treatment may be continued until disease progression or unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent prior to beginning protocol specific procedures
2. Histologically proven cancer at the first diagnosis. At study entry, it was desirable but not required to have histological or cytological proof of metastasis in the case of a 1 single metastatic target lesion.
3. Advanced neoplastic disease that was refractory to conventional treatment or for which no standard therapy existed
4. Progressive disease
5. Age 18-70 years
6. ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 2
7. Off previous anticancer (radio- or chemo-) therapy for at least 4 weeks and 6 weeks if prior nitrosoureas, mitomycin C; recovery from the toxic effects of prior treatment (Grade ≤1, except alopecia any grade)
8. Off previous immunotherapy for at least 1 week provided that patients did not have any residual signs of any toxicity
9. Adequate organ function including: neutrophils ≥2.0 × 109/L; platelets ≥100 × 109/L, creatinine <120 μmol/L (if borderline creatinine values, the creatinine clearance had to be ≥60 mL/min); total bilirubin within normal limit; alanine aminotransferase (ALT)/aspartate aminotransferase (AST)/alkaline phosphatase (ALP) ≤2.5-fold the upper normal limits of the institutional norms (ALP ≤2.5 UNL)
10. Patients registered in this trial had to be treated and followed at the participating centers
11. Patients who had received previous treatment with paclitaxel or docetaxel could be included provided that they did not have any residual signs of taxane toxicity (except alopecia any grade and peripheral neuropathy Grade 1)

Exclusion Criteria:

1. Hematological malignancies
2. Pregnant or lactating women or women of childbearing potential (eg, not using adequate contraception)
3. Symptomatic brain metastases
4. Previous extensive radiotherapy (>20% of bone marrow area)
5. Current peripheral neuropathy of any origin including significant residual symptoms due to the use of eg, vinca-alkaloids or platinum ≥Grade 2 according to the National Cancer Institute common terminology criteria for adverse events.
6. Other serious illness or medical conditions:

   * Congestive heart failure or angina pectoris even if medically controlled, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmias
   * Existence of significant neurological or psychiatric disorders including dementia or seizures
   * Active infection
   * Uncontrolled peptic ulcer, unstable diabetes mellitus, or other contraindications for the use of corticosteroids
7. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to patient registration
8. Concurrent treatment with any other anticancer therapy
9. Concomitant radiotherapy
10. Concomitant treatment with corticosteroids. However, patients receiving chronic treatment with corticosteroids (≤20 mg of methylprednisolone or ≤4 mg of dexamethasone or equivalent dose of other corticosteroids), for whatever reason, were eligible.
11. More than 2 prior chemotherapy regimens containing mitomycin C or nitrosoureas
12. More than 2 prior chemotherapy regimens for advanced disease
13. Prior history of severe allergic reaction to docetaxel or paclitaxel
14. Prior intensive chemotherapy with autologous stem cell rescue

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1999-10; Primary Completion 2002-08 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 35 months
Maximum tolerated dose | Up to 35 months

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to 35 months
Antitumor activity | Up to 35 months
  Measured by X-ray, ultrasound and/or scans
Pharmacokinetic parameters including Cmax, AUC(0-t), AUC, t, t1/2λz (h), Vss, CL, accumulation ratio, Tmax metabolite ratio and F (bioavailability) | Up to 35 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Sanofi, Paris, France
- Sanofi, Barcelona, Spain

REFERENCES:
- [Derived] Fumoleau P, Trigo JM, Isambert N, Semiond D, Gupta S, Campone M. Phase I dose-finding study of cabazitaxel administered weekly in patients with advanced solid tumours. BMC Cancer. 2013 Oct 7;13:460. doi: 10.1186/1471-2407-13-460. PMID 24099585